CLINICAL TRIAL: NCT04341831
Title: Does Teicoplanin Powder Use In Lumbar Instrumentation Surgery Reduce Surgical Site Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Murat Sarikas, Orthopaedics surgeon, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 70366045618
Record Dates: First submitted 2020-04-08; First posted 2020-04-10 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Disc Herniation; Scoliosis Lumbar Region; Lumbar Spondylolisthesis; Lumbar Disc Lesion
Keywords: Spine Surgery; Teicoplanin powder; Surgical site infection; Posterior lumbar instrumentation
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement; Spondylolisthesis; Surgical Wound Infection | interventions — Teicoplanin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): We will be added 200mg teicoplanin powder around instrument for each level.
  Interventions: Drug: Teicoplanin
- Group 2 (No Intervention): We will not used any antibiotic powder in this group.

INTERVENTIONS:
Drug: Teicoplanin — We will be used 200mg Teicoplanin powder for each level of instrument.Hemovac drains will be used in either group. The drains will remain closed for 6 hours post-operatively for teicoplanin powder penetration in a surgical site.
  Other Names: Targocid
  Arms: Group 1

SUMMARY:
Infection after spinal surgery is one of the serious complications. Spinal surgery infection can cause high morbidity, mortality, and costs. In spite of different prophylactic methods, up to 15% of infection appears after spinal surgery.

Vancomycin powder, which is one of the most applied methods, seems to be effective and inexpensive. However, vancomycin administration may be inconvenient in elderly participants with high comorbidity and especially kidney problems.

The investigators aimed to reduce the rate of infection in the post-op 90-day period by adding per-op Teicoplanin powder onto the implant in participants scheduled for lumbar posterior instrumentation.

DETAILED DESCRIPTION:
Study Design:

The investigators will start trial after our institution's Clinical Research Ethics Committee approval. The protocol conforms to CONSORT guidelines for parallel-group randomized trials and the protocol is designed to conform to the principles of the Declaration of Helsinki.

Participant :

A literature review revealed that the surgical site infection rates after posterior instrumentation to be around 13-15%. Being a non-inferiority trial, the investigators hypothesized that the 90-day surgical site infection rates after posterior lumbar instrumentation should not be more than 1%. In order to find the difference of 14.0% between the two groups statistically significant, the minimum number of subjects required in each group was determined to be 55. (Power of 80 % and significance level at 0.05). To account for missing data, the drop-out rate was set to 10% and therefore, a total of 60 participants will be randomized.

The investigators will be included participants with spinal stenosis, LDH(Lumbar Disc Hernia), degenerative scoliosis or spondylolisthesis who did not respond to conservative treatment and participants in whom operation will be planned in the only lumbar spine. The investigators will be excluded participants with a history of malignancy, systemic inflammatory disease, severe cardiac insufficiency, morbid obesity (>40 kg/m2 or 35 or more and experiencing obesity-related health conditions) and participants who had undergone spine surgery previously. An informed consent form will be obtained from all participants.

The schedule for randomization will be randomly generated using a computer before the initiation of the trial. Participants will randomly be assigned in a 1:1 ratio. The investigators planned our study as double-blinded. Neither participants nor assessors will know about randomization results. The outcome assessor will be blinded to group allocation and won't be involved in providing the interventions. The statistician performing the statistical analyses will be blinded to group allocation.

Surgical procedures:

All surgeries will be performed by one surgeon under general anesthesia. The investigators will be used rod and pedicle screws of the same brand in all participants (Tasarım Med, Turkey)- using a standard posterior midline approach. All participants will be given 2 g cefazolin for infection prophylaxis and 1 g tranexamic acid for blood loss prophylaxis intravenously 30 min before the incision. In group 1 Teicoplanin powder will be placed on the rod and pedicle screws. The investigators will be added 200mg. teicoplanin powder around the instrument for each level. Hemovac drains will be used in either group. The drains will remain closed for 6 hours post-operatively for teicoplanin powder penetration in a surgical site.

All participants will be undergoing the same post-op rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar spinal stenosis,
* LDH(Lumbar Disc Hernia)
* Lumbar degenerative scoliosis
* Lumbar spondylolisthesis

Exclusion Criteria:

* History of malignancy
* Systemic inflammatory disease
* Severe cardiac insufficiency
* Morbid obesity (>40 kg/m2 or 35 or more and experiencing obesity-related health conditions)
* History of lumbar spine surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 90 days
  Surgical site infection rates will be compared between two goups

CONTACTS AND LOCATIONS:
Overall Officials: Murat Sarıkaş, MD, Principal Investigator — Bezmialem Vakif University

IPD SHARING:
Plan to Share IPD: No